CLINICAL TRIAL: NCT04544631
Title: Active and Passive Virtual Reality Distraction for Pain Management During Pediatric Burn Dressing Changes
Brief Title: VR for Pediatric Burn Dressing Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Henry Xiang, Professor and Center Director, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB16-00444
Record Dates: First submitted 2020-09-01; First posted 2020-09-10 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pain; Burns
Keywords: Pediatrics; Burns; Pain; Virtual Reality
MeSH Terms: conditions — Pain; Burns

STUDY DESIGN:
Intervention Model Description: A prospective, three-group between subject randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers and nurses did not know the group assignment until immediately prior to intervention. Following the dressing change procedure, a second researcher, blinded to the group assignment, asked participants a post-assessment that included questions about child and guardian perceived pain and subjective VR experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active VR (Experimental): Participants in the active VR group played a virtual reality game entitled "Virtual River Cruise". In this game, an otter floats down a river on a boat and players activate snow-blowing statues along the shore by focusing on them. The statues will emit snow if they are correctly aimed at by the child, and a thermometer placed in the front of the boat shows decreased temperatures as more snowflakes are blown. As feedback to reinforce continued engagement, a scoreboard placed beside the thermometer will show children the number of statues he/she has activated. Additionally, as the temperature drops, snow and ice will start piling up on the boat and its surroundings, providing an enhanced "cooling" experience for pediatric burn patients. Children interact with the immersive virtual reality environment by tilting their head, minimizing potential interference with the dressing change procedure.
  Interventions: Other: Virtual reality game as adjunctive pain management tool
- Passive VR (Experimental): Participants in the passive VR group were immersed in the same virtual reality environment as the active VR group, without any interactions with the VR game.
  Interventions: Other: Virtual reality game as adjunctive pain management tool
- Standard Care Control (No Intervention): Participants in the standard group received routinely used distraction tools provided in the clinical setting, such as iPads, music, books, and/or talking.

INTERVENTIONS:
Other: Virtual reality game as adjunctive pain management tool — A smart phone virtual reality-based pain alleviation tool (VR-PAT).
  Arms: Active VR; Passive VR

SUMMARY:
This study evaluated a smart phone virtual reality (VR) to manage pediatric burn dressing pain. A randomized controlled trial was conducted among 90 patients (6-17 years). Active VR participants played the game, passive VR group were immersed in the same VR without interactions, and a standard care group served as the control. One researcher administered VR and observed pain while another researcher administered post-trial survey that measured child's perceived pain and VR experience. Nurses were asked to report the clinical utility.

ELIGIBILITY:
Inclusion Criteria:

* children age 6-17 years (inclusive)
* admitted or seen in the outpatient clinic for a burn injury
* spoke English as primary language

Exclusion Criteria:

* a severe burn on the face or head that prevented the utilization of the VR
* cognitive or motor impairment that prevented valid administration of study measures
* visual or hearing impairments that prevented interaction with the VR environment
* did not have a legal guardian present to give consent

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
Observed pain | During outpatient burn dressing change, on average lasting about 15 minutes.
  Researcher observed pain of patient based on the Face Legs Activity Cry and Consolability behavioral pain assessment tool (FLACC-r), using 0,1,2 numerical scale for category of face, legs, activity, cry, and consolability. Total scores range from 0-10 with higher scores indicating more pain.
Patient self-reported pain | During outpatient burn dressing change, on average lasting about 15 minutes.
  Patient-perceived pain using 0-100 scale Visual Analog Scales (VAS), 0(min)-100(max), higher score for worse outcome.

SECONDARY OUTCOMES:
VR experience self-reported by patient and parents | During outpatient burn dressing change, on average lasting about 15 minutes.
  Self-reported virtual reality experience using patient and parent survey questions (5-6 survey items) about their experience in using virtual reality during burn wound care. Questions are a mixture of yes/no and a 100 Visual Analog Scale (VAS) with 0 being "Not at All" and 100 being "Very Much"
Simulator sickness symptoms of patient | During outpatient burn dressing change, on average lasting about 15 minutes.
  Simulator sickness symptoms using the Simulator Sickness Questionnaire (SSQ), which has 15 survey items with possible choices of "None", "Slight", "Moderate", and "Severe".
Nurse reported feasibility of VR in clinical burn wound care | During outpatient burn dressing change, on average lasting about 15 minutes.
  Attending nurse answered two questions using a survey questionnaire about clinical feasibility of VR using scale ranging from "not at all" to "very easy".

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiang, MD, MPH, PhD, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No
IPD are confidential patient data so we are not allowed to share the data with other researchers

REFERENCES:
- [Result] Xiang H, Shen J, Wheeler KK, Patterson J, Lever K, Armstrong M, Shi J, Thakkar RK, Groner JI, Noffsinger D, Giles SA, Fabia RB. Efficacy of Smartphone Active and Passive Virtual Reality Distraction vs Standard Care on Burn Pain Among Pediatric Patients: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jun 1;4(6):e2112082. doi: 10.1001/jamanetworkopen.2021.12082. PMID 34152420
- [Result] Vest E, Armstrong M, Olbrecht VA, Thakkar RK, Fabia RB, Groner JI, Noffsinger D, Tram NK, Xiang H. Association of Pre-procedural Anxiety With Procedure-Related Pain During Outpatient Pediatric Burn Care: A Pilot Study. J Burn Care Res. 2023 May 2;44(3):610-617. doi: 10.1093/jbcr/irac108. PMID 35913793
- [Result] Jain S, Armstrong M, Luna J, Thakkar RK, Fabia R, Groner JI, Noffsinger D, Ni A, Nelson E, Xiang H. Features of virtual reality impact effectiveness of VR pain alleviation therapeutics in pediatric burn patients: A randomized clinical trial. PLOS Digit Health. 2024 Jan 25;3(1):e0000440. doi: 10.1371/journal.pdig.0000440. eCollection 2024 Jan. PMID 38271320
- [Result] Jones K, Armstrong M, Luna J, Thakkar RK, Fabia R, Groner JI, Noffsinger D, Ni A, Griffin B, Xiang H. Age and Sex Differences of Virtual Reality Pain Alleviation Therapeutic During Pediatric Burn Care: A Randomized Clinical Trial. J Med Ext Real. 2024 Jul 24;1(1):163-173. doi: 10.1089/jmxr.2024.0004. eCollection 2024 Jul. PMID 39091668